CLINICAL TRIAL: NCT06349161
Title: Long-term Outcome of Retroperitoneoscopic One-trocar-assisted Pyeloplasty: A Single-center and Single-surgeon Experience
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Nguyen Thanh Quang, Pediatric Surgeon, National Children's Hospital, Vietnam
Other Study IDs: 1451_02/BVNTW-VNCSKTE
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Ureteropelvic Junction Obstruction
Keywords: Hydronephrosis; Laparoscopic; Pyeloplasty; Minimally invasive; Ureteropelvic junction obstruction
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral; Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ureteropelvic junction obstruction: UPJO with severe hydronephrosis, with or without parenchymal atrophy (Society for Fetal Urology grade III or IV), recurrent urinary tract infections (UTI), prolonged drainage parameters with T1/2 > 20 minutes, and/or differential renal function (DRF) less than 40%.
  Interventions: Procedure: One-trocar-assisted pyeloplasty

INTERVENTIONS:
Procedure: One-trocar-assisted pyeloplasty — Positioned in a full lateral decubitus posture. A 12mm incision was made below the 12th rib, followed by a muscle-sparing technique to access and open the Gerota's fascia. A 10mm balloon trocar was inserted, and CO2 was insufflated to a pressure of 12 mmHg at a flow rate of 3L. An operative scope with dual channels was introduced for retroperitoneal dissection, utilizing a peanut to expand the working space. The proximal ureter, UPJ, and renal pelvis were visualized, and the UPJ was mobilized and exteriorized under direct visualization to prevent torsion. Anderson-Hynes dismembered pyeloplasty was performed using a 6/0 PDS suture, with possible enlargement of the incision if necessary. A 4 French double J ureteral stent was inserted antegradely before completing the anastomosis, verified by methylene blue presence at the anastomotic site. A final retroperitoneoscopic assessment ensured proper alignment of the anastomosis, with closure of the incision site without drain placement.

SUMMARY:
Open surgical dismembered pyeloplasty has traditionally been the preferred method for treating ureteropelvic junction obstruction (UPJO), with a success rate exceeding 94%. However, it is associated with drawbacks such as increased postoperative pain, extended hospital stays, and visible scarring. Minimally invasive alternatives, including laparoscopic pyeloplasty (LP) and robot-assisted laparoscopic pyeloplasty (RALP), have gained popularity since their introduction in 1993, offering comparable success rates to open surgery while providing cosmetic benefits and shorter hospital stays. Nevertheless, these techniques present challenges in pediatric patients, including limited working space, technical complexities, and prolonged operative times. The retroperitoneoscopic one-trocar-assisted pyeloplasty (OTAP) method, introduced in 2007, combines the advantages of minimally invasive surgery with the success rates of standard dismembered pyeloplasty. Despite favorable outcomes reported by several researchers, comprehensive studies regarding long-term follow-up and clinical outcomes are lacking. This study aims to evaluate the long-term outcomes of OTAP, addressing this gap in the medical literature.

DETAILED DESCRIPTION:
Open surgical dismembered pyeloplasty has historically been the gold standard for managing ureteropelvic junction obstruction (UPJO), boasting a success rate exceeding 94%. However, the requisite incision and muscle dissection can lead to increased postoperative pain, prolonged hospitalization, and undesirable scarring. In recent decades, there has been a growing interest in minimally invasive pyeloplasty, commencing with its inception in 1993. Laparoscopic pyeloplasty (LP) and robot-assisted laparoscopic pyeloplasty (RALP) have emerged as widely embraced and dependable therapeutic modalities for UPJO. Both techniques have demonstrated success rates comparable to those of open pyeloplasty while conferring advantages in terms of cosmetic outcomes and length of hospital stay.

However, despite their merits, minimally invasive approaches pose certain limitations in pediatric patients, including restricted working space, technical intricacies, prolonged operative time, steep learning curves, and the need for expensive instrumentation. Conventional laparoscopic pyeloplasty has encountered slow uptake due to its technical demands and substantial learning curve. The evolution of RALP over the past decade appears to mitigate the learning curve associated with intracorporeal suturing and anastomosis time. Nonetheless, RALP necessitates three to four port placements and a sizeable initial financial investment.

In 2007, Lima et al. introduced the retroperitoneoscopic one-trocar-assisted pyeloplasty (OTAP) approach, which "combines the advantages of a minimally invasive technique with the high success rate of standard dismembered pyeloplasty". Several other researchers have replicated this technique with favorable outcomes. Nevertheless, a dearth of comprehensive studies delineating long-term follow-up and clinical outcomes persists in the medical literature. The aim of this study is to evaluate the long-term outcomes of OTAP.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 months to 5 years old with UPJ obstruction who underwent OTAP between May 2011 and June 2013.
* Anteroposterior renal pelvic diameter of 20 mm or greater, which demonstrated progressive enlargement on subsequent ultrasounds, coupled with impaired split renal function of 40% or less on nuclear scan, characterized by a T1/2 > 20 minutes
* The surgical technique performed must be one trocar-assisted pyeloplasty

Exclusion Criteria:

* A history of previous renal surgery
* UPJO associated with other urinary tract anomalies
* Identification of crossing lower pole renal vessels as the cause of obstruction.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The cohort comprised seventy pediatric patients who underwent RALP for UPJO at the National Hospital of Pediatrics between May 2011 and June 2013. Preoperative diagnostic evaluations included blood tests, urinalysis, urine culture, renal ultrasonography (US), voiding cystourethrogram (VCUG) to exclude vesicoureteral reflux disease, magnetic resonance imaging (MRI) to exclude other associated renal pathologies, and technetium-99m diethylenetriamine penta-acetic acid (99mTc DTPA) scans.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
Operative time | through study completion (3 years)
  The average and range of operative time (minutes) using the OTAP technique
Conversion to open | through study completion (3 years)
  Incidence in which the operation must be switch to open surgery
Extension of skin incision | through study completion (3 years)
  Incidence in which the original incision of the skin must be extended to accommodate UPJ mobilization
Postoperative complications | through study completion (3 years)
  Complications after OTAP including febrile UTI
Median length of hospital stays | through study completion (3 years)
  The average time (days) the patient stays at the hospital post-operation
Median follow up length | through study completion (3 years)
  The average time (months) the patient revisit the hospital for follow-up sessions
Post-operative mean APD | through study completion (3 years)
  The average anterior posterior diameter (mm) of the renal pelvis post-operation
Post-operative mean DRF | through study completion (3 years)
  The average different renal function (%) (measurement of each kidney's ability to extract tracer from blood) after the operation
Mean incision length | through study completion (3 years)
  The average length (mm) of the primary incision during the operation
Recurrence | through study completion (3 years)
  Instances of symptoms reappeared after the completion of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Quang T Nguyen, M.D., Principal Investigator — : Department of Pediatric Surgery, The National Hospital of Pediatrics, Hanoi, Vietnam
Locations (1):
- The National Hospital of Pediatrics, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ANDERSON JC, HYNES W. Retrocaval ureter; a case diagnosed pre-operatively and treated successfully by a plastic operation. Br J Urol. 1949 Sep;21(3):209-14. doi: 10.1111/j.1464-410x.1949.tb10773.x. No abstract available. PMID 18148283
- [Background] Mikkelsen SS, Rasmussen BS, Jensen TM, Hanghoj-Petersen W, Christensen PO. Long-term follow-up of patients with hydronephrosis treated by Anderson-Hynes pyeloplasty. Br J Urol. 1992 Aug;70(2):121-4. doi: 10.1111/j.1464-410x.1992.tb15688.x. PMID 1393432
- [Background] Schuessler WW, Grune MT, Tecuanhuey LV, Preminger GM. Laparoscopic dismembered pyeloplasty. J Urol. 1993 Dec;150(6):1795-9. doi: 10.1016/s0022-5347(17)35898-6. PMID 8230507
- [Background] Inagaki T, Rha KH, Ong AM, Kavoussi LR, Jarrett TW. Laparoscopic pyeloplasty: current status. BJU Int. 2005 Mar;95 Suppl 2:102-5. doi: 10.1111/j.1464-410X.2005.05208.x. PMID 15720343
- [Background] Braga LH, Lorenzo AJ, Bagli DJ, Mahdi M, Salle JL, Khoury AE, Farhat WA. Comparison of flank, dorsal lumbotomy and laparoscopic approaches for dismembered pyeloplasty in children older than 3 years with ureteropelvic junction obstruction. J Urol. 2010 Jan;183(1):306-11. doi: 10.1016/j.juro.2009.09.008. PMID 19914659
- [Background] Sweeney DD, Ost MC, Schneck FX, Docimo SG. Laparoscopic pyeloplasty for ureteropelvic junction obstruction in children. J Laparoendosc Adv Surg Tech A. 2011 Apr;21(3):261-5. doi: 10.1089/lap.2010.0155. Epub 2011 Feb 1. PMID 21284513
- [Background] Piaggio LA, Franc-Guimond J, Noh PH, Wehry M, Figueroa TE, Barthold J, Gonzalez R. Transperitoneal laparoscopic pyeloplasty for primary repair of ureteropelvic junction obstruction in infants and children: comparison with open surgery. J Urol. 2007 Oct;178(4 Pt 2):1579-83. doi: 10.1016/j.juro.2007.03.159. Epub 2007 Aug 16. PMID 17707047
- [Background] Hemal AK, Goel R, Goel A. Cost-effective laparoscopic pyeloplasty: single center experience. Int J Urol. 2003 Nov;10(11):563-8. doi: 10.1046/j.1442-2042.2003.00706.x. PMID 14633078
- [Background] Boysen WR, Gundeti MS. Robot-assisted laparoscopic pyeloplasty in the pediatric population: a review of technique, outcomes, complications, and special considerations in infants. Pediatr Surg Int. 2017 Sep;33(9):925-935. doi: 10.1007/s00383-017-4082-7. Epub 2017 Apr 1. PMID 28365863
- [Background] Passerotti CC, Passerotti AM, Dall'Oglio MF, Leite KR, Nunes RL, Srougi M, Retik AB, Nguyen HT. Comparing the quality of the suture anastomosis and the learning curves associated with performing open, freehand, and robotic-assisted laparoscopic pyeloplasty in a swine animal model. J Am Coll Surg. 2009 Apr;208(4):576-86. doi: 10.1016/j.jamcollsurg.2009.01.010. PMID 19476793
- [Background] Howe A, Kozel Z, Palmer L. Robotic surgery in pediatric urology. Asian J Urol. 2017 Jan;4(1):55-67. doi: 10.1016/j.ajur.2016.06.002. Epub 2016 Sep 6. PMID 29264208
- [Background] Song SH, Lee C, Jung J, Kim SJ, Park S, Park H, Kim KS. A comparative study of pediatric open pyeloplasty, laparoscopy-assisted extracorporeal pyeloplasty, and robot-assisted laparoscopic pyeloplasty. PLoS One. 2017 Apr 20;12(4):e0175026. doi: 10.1371/journal.pone.0175026. eCollection 2017. PMID 28426695
- [Background] Monn MF, Bahler CD, Schneider EB, Whittam BM, Misseri R, Rink RC, Sundaram CP. Trends in robot-assisted laparoscopic pyeloplasty in pediatric patients. Urology. 2013 Jun;81(6):1336-41. doi: 10.1016/j.urology.2013.01.025. Epub 2013 Mar 19. PMID 23522294
- [Background] Lima M, Tursini S, Ruggeri G, Gargano T, Libri M, Domini M. One trocar assisted pyeloplasty (OTAP): initial experience and codification of a technique. Pediatr Med Chir. 2007 Mar-Apr;29(2):108-11. PMID 17461099
- [Background] Mei H, Pu J, Yang C, Zhang H, Zheng L, Tong Q. Laparoscopic versus open pyeloplasty for ureteropelvic junction obstruction in children: a systematic review and meta-analysis. J Endourol. 2011 May;25(5):727-36. doi: 10.1089/end.2010.0544. Epub 2011 Apr 8. PMID 21476861
- [Background] Huang Y, Wu Y, Shan W, Zeng L, Huang L. An updated meta-analysis of laparoscopic versus open pyeloplasty for ureteropelvic junction obstruction in children. Int J Clin Exp Med. 2015 Apr 15;8(4):4922-31. eCollection 2015. PMID 26131065
- [Background] Andolfi C, Adamic B, Oommen J, Gundeti MS. Robot-assisted laparoscopic pyeloplasty in infants and children: is it superior to conventional laparoscopy? World J Urol. 2020 Aug;38(8):1827-1833. doi: 10.1007/s00345-019-02943-z. Epub 2019 Sep 10. PMID 31506749
- [Result] Minnillo BJ, Cruz JA, Sayao RH, Passerotti CC, Houck CS, Meier PM, Borer JG, Diamond DA, Retik AB, Nguyen HT. Long-term experience and outcomes of robotic assisted laparoscopic pyeloplasty in children and young adults. J Urol. 2011 Apr;185(4):1455-60. doi: 10.1016/j.juro.2010.11.056. Epub 2011 Feb 19. PMID 21334663
- [Result] Blanc T, Kohaut J, Elie C, Clermidi P, Pio L, Harte C, Bronnimann E, Botto N, Rousseau V, Sonigo P, Vaessen C, Lottmann H, Aigrain Y. Retroperitoneal Approach for Ureteropelvic Junction Obstruction: Encouraging Preliminary Results With Robot-Assisted Laparoscopic Repair. Front Pediatr. 2019 May 28;7:209. doi: 10.3389/fped.2019.00209. eCollection 2019. PMID 31192176
- [Result] Caione P, Lais A, Nappo SG. One-port retroperitoneoscopic assisted pyeloplasty versus open dismembered pyeloplasty in young children: preliminary experience. J Urol. 2010 Nov;184(5):2109-15. doi: 10.1016/j.juro.2010.06.126. Epub 2010 Sep 18. PMID 20851429
- [Result] Chen WC, Huang SY, Yeh CM, Chou CM. Hybrid Retroperitoneoscopic Pyeloplasty for Congenital Ureteropelvic Junction Obstruction in Infants Weighing Less than 10 kg. J Laparoendosc Adv Surg Tech A. 2021 Jul;31(7):843-848. doi: 10.1089/lap.2020.0799. Epub 2021 May 27. PMID 34042526
- [Result] Lima M, Ruggeri G, Messina P, Tursini S, Destro F, Mogiatti M. One-trocar-assisted pyeloplasty in children: an 8-year single institution experience. Eur J Pediatr Surg. 2015 Jun;25(3):262-8. doi: 10.1055/s-0034-1372459. Epub 2014 Apr 4. PMID 24705997
- [Result] Bajpai M, Khanna K, Khanna V, Goel P, Baidya DK. Lumboscopic-Assisted Pyeloplasty: A Single-Port, Retroperitoneoscopic Approach for Children with Pelvi-Ureteric Junction Obstruction. J Indian Assoc Pediatr Surg. 2020 May-Jun;25(3):163-168. doi: 10.4103/jiaps.JIAPS_5_19. Epub 2020 Apr 11. PMID 32581444
- [Result] Chen Z, Chen X, Wu ZH, Luo YC, He Y, Li NN, Xie CQ, Lai C. Feasibility and safety of retroperitoneal laparoendoscopic single-site dismembered pyeloplasty: a clinical report of 10 cases. J Laparoendosc Adv Surg Tech A. 2012 Sep;22(7):685-90. doi: 10.1089/lap.2012.0164. Epub 2012 Jul 30. PMID 22845552
- [Result] Alizadeh F, Haghdani S, Seydmohammadi B. Minimally invasive open pyeloplasty in children: Long-term follow-up. Turk J Urol. 2020 Sep;46(5):393-397. doi: 10.5152/tud.2020.20011. Epub 2020 May 21. PMID 32449670
- [Result] He Y, Song H, Liu P, Sun N, Tian J, Li M, Li N, Qu Y, Han W, Feng G, Ni X, Zhang W. Primary laparoscopic pyeloplasty in children: A single-center experience of 279 patients and analysis of possible factors affecting complications. J Pediatr Urol. 2020 Jun;16(3):331.e1-331.e11. doi: 10.1016/j.jpurol.2020.03.028. Epub 2020 Apr 10. PMID 32334969
- [Result] Scuderi MG, Arena S, Di Benedetto V. One-trocar-assisted pyeloplasty. J Laparoendosc Adv Surg Tech A. 2011 Sep;21(7):651-4. doi: 10.1089/lap.2010.0115. Epub 2011 Jul 21. PMID 21777059
- [Derived] Nguyen QT, Nguyen TM, Le DA, Nguyen LVM, Dang TT, Nguyen SH, Nguyen VHK, Nguyen LT. Long-term outcome of retroperitoneoscopic one-trocar-assisted pyeloplasty: a single-center and single-surgeon experience. Int Urol Nephrol. 2024 Nov;56(11):3469-3477. doi: 10.1007/s11255-024-04091-9. Epub 2024 May 27. PMID 38797767